CLINICAL TRIAL: NCT03038204
Title: The Papillary Muscle Approximation Provide Stability of Mitral Valve Repair for Ischemic Mitral Regurgitation
Acronym: PMA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Federal Centre of Cardiovascular Surgery, Russia (Other)
Responsible Party: Principal Investigator, Mikulyak Artur, Principal Investigator, Cardiovascular surgeon, The Federal Centre of Cardiovascular Surgery, Russia
Other Study IDs: FederalCCS 001
Record Dates: First submitted 2017-01-16; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Mitral Regurgitation
Keywords: Papillary muscles approximation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PMA+MVA+CABG: patients with ischemic cardiomyopathy and mitral regurgitation who underwent coronary artery bypass grafting, mitral annuloplasty, and papillary muscles approximation.
  Interventions: Procedure: The papillary muscle approximation
- MVA+CABG: patients with ischemic cardiomyopathy who underwent coronary artery bypass grafting and mitral valve annuloplasty.

INTERVENTIONS:
Procedure: The papillary muscle approximation — Surgery is performed through median sternotomy, aortic and bicaval cannulation, normothermic perfusion, and antegrade cardioplegia with the use of cardioplegic solution.
  After coronary anastomosis, the mitral valve is exposed by a transseptal incision.
  The papillary muscles are approximated through the mitral valve at the level of papillary muscles heads. Nonabsorbable, braided sutures of 2-0 (Ethibond, Ethicon, Inc.) with PTFE felt pledgets are used for this purpose.
  Annuloplasty mitral rings of different sizes are anchored using multiple deep U-shaped stitches of Ethibond 2-0 (Ethicon, Inc., USA). After MV repair, the LV is forcefully filled with saline water to test the valve competence. After satisfactory hydraulic test walls of the heart chambers are sutured.
  Groups: PMA+MVA+CABG

SUMMARY:
Recent publications show that an adjunctive subvalvular repair during mitral annuloplasty for secondary mitral regurgitation effective in preventing recurrent regurgitation. One of these procedures is the papillary muscles approximation. However, the safety and the positive impact of this method are still in doubt.

DETAILED DESCRIPTION:
Ischemic mitral regurgitation develops in 10-50% of patients after myocardial infarction. Among several surgical procedures, mitral ring annuloplasty has been the method of choice for a considerable period. However, mitral regurgitation recurrence after surgery has a reported occurrence that ranges from 5% to 58%. Careful consideration of the mechanisms underlying recurrence of mitral regurgitation after annuloplasty might explain the unsatisfactory outcomes. The pathophysiology of IMR is complex and results from the imbalance between closing and tethering forces acting on the mitral valve. Enlargement of the left ventricular chamber, and displacement of papillary muscles in apical and lateral direction increase the tethering forces. Left ventricular and papillary muscle dyssynchrony, reduced myocardial contractility decrease closing forces, which lead to impaired leaflet coaptation and appearance of mitral regurgitation. Thus, treatment of mitral insufficiency requires an integrated approach affecting all units of the pathogenesis of MR recurrence.

Recent publications show that an adjunctive subvalvular repair during mitral annuloplasty for secondary mitral regurgitation effective in preventing recurrent regurgitation. One of these procedures is the papillary muscles approximation. However, the safety and the positive impact of this method are still in doubt. This study is conducted to identify the positive qualities and safety of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic cardiomyopathy,
* Ischemic mitral regurgitation.

Exclusion Criteria:

* Degenerative mitral valve disease,
* Unstable angina,
* Recent myocardial infarction (< 6 months),
* Papillary muscles rupture,
* Severe right ventricular dysfunction,
* Multiple organ failures,
* Concomitant left ventricular reconstruction,
* Aortic valve procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with ischemic cardiomyopathy and coexisting IMR were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Mitral regurgitation severity (1,2 or 3) | 1 year
  Mitral regurgitation severity is the main indicator of the effectiveness of mitral valve plasty. Evaluation of mitral regurgitation was performed in accordance with the recommendations of the American Society of Echocardiography (ASE). Recurrence of mitral regurgitation 2 and more was considered as significant.

SECONDARY OUTCOMES:
End-diastolic volume (ml), end-systolic volume (ml), stroke volume (ml) | 1 year
  Assessment of left ventricular dimensions.
Ejection fraction (%) | 1 year
  Assessment of myocardial contractility.
Systolic interpapillary muscle distance (mm), diastolic interpapillary muscle distance (mm), coaptation depth (mm), coaptation length (mm) | 1 year
  Assessment of the impact of the surgery on the mitral valve configuration.
Tenting area (mm^2) | 1 year
  Assessment of the impact of the surgery on the configuration of the mitral valve.

OTHER OUTCOMES:
Age (years) | 1 year
  Description and comparison of groups of patients
Body mass index (kg/m^2) | 1 year
  Description and comparison of groups of patients.
Body surface area (m^2) | 1 year
  Description and comparison of groups of patients.
NYHA (I, II, III or IV) | 1 year
  Description and comparison of groups of patients.
EuroSCORE | 1 year
  Description and comparison of groups of patients.
Six minute walk test (m) | 1 year
  Description and comparison of groups of patients.
Hypertension (absence, stage 1, 2 or 3) | 1 year
  Description and comparison of groups of patients. Impact of the factor on the long-term survival.
Diabetes mellitus (absence, insulin-dependent or noninsulin-dependent) | 1 year
  Description and comparison of groups of patients. Impact of the factor on the long-term survival.
Obesity (absence, class 1, 2 or 3) | 1 year
  Description and comparison of groups of patients. Impact of the factor on the long-term survival.
Multifocal atherosclerosis (presence or absence) | 1 year
  Description and comparison of groups of patients. Impact of the factor on the long-term survival.
COPD (absence, GOLD 1, 2, 3 or 4) | 1 year
  Description and comparison of groups of patients. Impact of the factor on the long-term survival.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Manabe S, Shimokawa T, Fukui T, Tabata M, Takanashi S. Impact of papillary muscle approximation on mitral valve configuration in the surgical correction of ischemic mitral regurgitation. Thorac Cardiovasc Surg. 2012 Jun;60(4):269-74. doi: 10.1055/s-0032-1304536. Epub 2012 May 1. PMID 22549757
- [Result] Roshanali F, Vedadian A, Shoar S, Naderan M, Mandegar MH. Efficacy of papillary muscle approximation in preventing functional mitral regurgitation recurrence in high-risk patients with ischaemic cardiomyopathy and mitral regurgitation. Acta Cardiol. 2013 Jun;68(3):271-8. doi: 10.1080/ac.68.3.2983421. PMID 23882872
- [Result] Kron IL, Hung J, Overbey JR, Bouchard D, Gelijns AC, Moskowitz AJ, Voisine P, O'Gara PT, Argenziano M, Michler RE, Gillinov M, Puskas JD, Gammie JS, Mack MJ, Smith PK, Sai-Sudhakar C, Gardner TJ, Ailawadi G, Zeng X, O'Sullivan K, Parides MK, Swayze R, Thourani V, Rose EA, Perrault LP, Acker MA; CTSN Investigators. Predicting recurrent mitral regurgitation after mitral valve repair for severe ischemic mitral regurgitation. J Thorac Cardiovasc Surg. 2015 Mar;149(3):752-61.e1. doi: 10.1016/j.jtcvs.2014.10.120. Epub 2014 Nov 6. PMID 25500293
- [Result] Rama A, Praschker L, Barreda E, Gandjbakhch I. Papillary muscle approximation for functional ischemic mitral regurgitation. Ann Thorac Surg. 2007 Dec;84(6):2130-1. doi: 10.1016/j.athoracsur.2007.04.056. PMID 18036963
- [Result] Ishikawa S, Ueda K, Kawasaki A, Neya K, Suzuki H. Papillary muscle sandwich plasty for ischemic mitral regurgitation: a new simple technique. J Thorac Cardiovasc Surg. 2008 Jun;135(6):1384-6. doi: 10.1016/j.jtcvs.2007.12.034. No abstract available. PMID 18544392
- [Result] Yamaguchi A, Adachi K, Yuri K, Kimura N, Kimura C, Tamura A, Adachi H. Reduction of mitral valve leaflet tethering by procedures targeting the subvalvular apparatus in addition to mitral annuloplasty. Circ J. 2013;77(6):1461-5. doi: 10.1253/circj.cj-12-1148. Epub 2013 Feb 20. PMID 23428660
- [Result] Wakasa S, Kubota S, Shingu Y, Ooka T, Tachibana T, Matsui Y. The extent of papillary muscle approximation affects mortality and durability of mitral valve repair for ischemic mitral regurgitation. J Cardiothorac Surg. 2014 Jun 3;9:98. doi: 10.1186/1749-8090-9-98. PMID 24893928